CLINICAL TRIAL: NCT02305888
Title: Safety of LEO 43204 0.018%, 0.037% and 0.1% for Actinic Keratosis Applied Once Daily for Three Consecutive Days on Face/Chest, Scalp and Trunk/Extremities, Respectively
Brief Title: Safety of LEO 43204 for Actinic Keratosis Applied on Face/Chest, Scalp and Trunk/Extremities, Respectively
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP0084-1148
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2019-02

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — LEO 43204

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LEO 43204, 0.018% once daily for 3 days (Experimental)
  Interventions: Drug: LEO 43204
- LEO 43204, 0.037% once daily for 3 days (Experimental)
  Interventions: Drug: LEO 43204
- LEO 43204, 0.1% once daily for 3 days (Experimental)
  Interventions: Drug: LEO 43204

INTERVENTIONS:
Drug: LEO 43204 — Treatment of actinic keratosis

SUMMARY:
The objective of the trial is to investigate the Safety of LEO 43204 0.018%, 0.037% and 0.1% for actinic keratosis applied once daily for three consecutive days on face/chest, scalp and trunk/extremities, respectively.

ELIGIBILITY:
Inclusion Criteria:

Subjects with 5 to 20 clinically typical, visible and, discrete, nonhyperkeratotic and non-hypertrophic AKs within a selected treatment area of sun-damaged skin on either:

* The full face
* The full balding scalp
* A contiguous area of approximately 250 cm2 on trunk or extremities

Exclusion Criteria:

Location of the treatment area (full face, full balding scalp or chest) within 5 cm of an incompletely healed wound or within 5 cm of a suspected basal cell carcinoma (BCC) or SCC.

Previously assigned treatment in this clinical trial or previously participated in a clinical trial in the LEO 43204 programme.

Treatment with ingenol mebutate gel in the selected treatment area within the last 12 months

Lesions in the treatment area that have: atypical clinical appearance (e.g. cutaneous horns) and/or, recalcitrant disease (e.g., did not respond to cryotherapy on two previous occasions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Siegel, MD, Principal Investigator — Long Island Skin Cancer and Dermatologic Surgery
Locations (1):
- Long Island Skin Cancer and Dermatologic Surgery, Smithtown, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siegel DM, Tyring S, Nahm WK, Osterdal ML, Petersen AH, Berman B. Three-day Field Treatment with Ingenol Disoxate (LEO 43204) for Actinic Keratosis: A Phase II Trial. J Clin Aesthet Dermatol. 2017 Dec;10(12):19-26. Epub 2017 Dec 1. PMID 29399263
- [Derived] Berman B, Tyring S, Nahm WK, Osterdal ML, Petersen AH, Siegel DM. Three-Day Field Treatment with Ingenol Disoxate (LEO 43204) for Actinic Keratosis: Cosmetic Outcomes and Patient Satisfaction from a Phase II Trial. J Clin Aesthet Dermatol. 2017 Nov;10(11):26-32. Epub 2017 Nov 1. PMID 29399258
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Groups:
- LEO 43204 0.018% Face/Chest: Treatment with LEO 43204 0.018% gel once daily for 3 consecutive days on the full face or a contiguous area on the chest of approximately 250 cm2.
- LEO 43204 0.037% Scalp: Treatment with LEO 43204 0.037% gel once daily for 3 consecutive days on the full balding scalp of an area greater than 25 cm2 and up to approximately 250 cm2.
- LEO 43204 0.1% Trunk/Extremities: Treatment with LEO 43204 0.1% gel once daily for 3 consecutive days on a contiguous area of approximately 250 cm2 on trunk or extremities (excluding chest).
Period: Overall Study
Arm/Group | LEO 43204 0.018% Face/Chest | LEO 43204 0.037% Scalp | LEO 43204 0.1% Trunk/Extremities
Started | 63 | 63 | 63
Completed | 63 | 62 | 62
Not Completed | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population was based on the full analysis set, defined as all participants who assigned to treatment and who met the inclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | LEO 43204 0.018% Face/Chest | LEO 43204 0.037% Scalp | LEO 43204 0.1% Trunk/Extremities | Total
Number analyzed (Participants) | 63 | 63 | 62 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (8.8) | 67.7 (9.6) | 66.7 (9.6) | 66.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 1 | 23 | 47
  Male | 40 | 62 | 39 | 141
Region of Enrollment [Number; unit: participants]
  United States | 63 | 63 | 62 | 188

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing DLTs (Dose Limiting Toxicities) Based on LSRs (Local Skin Reactions)
Description: For face/chest, a DLT was defined as one or more of the following three LSRs:
  * Crusting Grade 4
  * Erosion/Ulceration Grade 4
  * Vesiculation/Pustulation Grade 4
  Or two or more of the following five LSRs:
  * Erythema Grade 4
  * Crusting Grade 3
  * Swelling Grade 4
  * Erosion/Ulceration Grade 3
  * Vesiculation/Pustulation Grade 3
  For scalp a DLT was defined as erosion/ulceration Grade 4
  For trunk/extremities a DLT was defined as one or more of the following three LSRs:
  * Crusting Grade 4
  * Erosion/Ulceration Grade 4
  * Vesiculation/Pustulation Grade 4
  Or two or more of the following four LSRs:
  * Crusting Grade 3
  * Swelling Grade 4
  * Erosion/Ulceration Grade 3
  * Vesiculation/Pustulation Grade 3
Time Frame: 8 days / From baseline (Day 1) to Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 43204 0.018% Face/Chest | LEO 43204 0.037% Scalp | LEO 43204 0.1% Trunk/Extremities
Number analyzed (Participants) | 63 | 63 | 62
Participants | 9 | 0 | 11

2. Secondary Outcome: Percent Reduction in AK Count Excluding Lesions Identified at Baseline as Hypertrophic/Hyperkeratotic
Description: The number of clinically visible actinic keratosis lesions (AKs) identified in the treatment area was recorded at baseline (Day 1), Week 4, and Week 8. This analysis excluded lesions identified at baseline as hypertrophic/hyperkeratotic.
Time Frame: 4 weeks and 8 weeks / From baseline to Week 4, and Week 8
Measure: Mean (95% Confidence Interval); unit: percentage of reduction
Arm/Group | LEO 43204 0.018% Face/Chest | LEO 43204 0.037% Scalp | LEO 43204 0.1% Trunk/Extremities
Number analyzed (Participants) | 63 | 63 | 62
percentage of reduction
  Week 4 | 81.2 [74.7 to 86.1] | 78.8 [71.6 to 84.1] | 59.0 [50.0 to 66.3]
  Week 8 | 78.9 [70.9 to 84.7] | 76.3 [66.7 to 83.1] | 69.1 [60.3 to 76.0]

3. Secondary Outcome: Percent Reduction in AK Count of Lesions Identified at Baseline as Hypertrophic/Hyperkeratotic
Description: Hypertrophic/Hyperkeratotic lesions were identified at baseline (Day 1), Week 4 and Week 8.
Time Frame: 4 weeks and 8 weeks / From baseline to Week 4, and Week 8
Population: For this efficacy analysis only participants with lesions identified as hypertrophic/hyperkeratotic at baseline were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: percentage of reduction
Arm/Group | LEO 43204 0.018% Face/Chest | LEO 43204 0.037% Scalp | LEO 43204 0.1% Trunk/Extremities
Number analyzed (Participants) | 9 | 10 | 16
percentage of reduction
  Week 4 | 78.7 [38.7 to 92.6] | 58.1 [6.8 to 81.2] | 36.0 [1.3 to 58.5]
  Week 8 | 68.5 [4.5 to 89.6] | 62.5 [-13.2 to 87.5] | 39.2 [7.9 to 59.9]

4. Secondary Outcome: Percentage of Participants With Complete Clearance of AKs
Description: Complete clearance was defined as no clinically visible AKs. This analysis excluded lesions identified at baseline as hypertrophic/hyperkeratotic.
Time Frame: 8 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LEO 43204 0.018% Face/Chest | LEO 43204 0.037% Scalp | LEO 43204 0.1% Trunk/Extremities
Number analyzed (Participants) | 63 | 63 | 62
percentage of participants | 36.5 [24.7 to 49.6] | 39.7 [27.6 to 52.8] | 22.6 [12.9 to 35.0]

ADVERSE EVENTS:
Time Frame: From baseline to Week 8±7 days
Arm/Group | LEO 43204 0.018% Face/Chest | LEO 43204 0.037% Scalp | LEO 43204 0.1% Trunk/Extremities
Serious Adverse Events (participants affected / at risk) | 1/63 | 0/63 | 0/62
Other Adverse Events (participants affected / at risk) | 35/63 | 47/63 | 43/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LEO 43204 0.018% Face/Chest (N=63) | LEO 43204 0.037% Scalp (N=63) | LEO 43204 0.1% Trunk/Extremities (N=62)
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LEO 43204 0.018% Face/Chest (N=63) | LEO 43204 0.037% Scalp (N=63) | LEO 43204 0.1% Trunk/Extremities (N=62)
Application site pain (General disorders) | 28 | 34 | 26
Application site pruritus (General disorders) | 18 | 23 | 21
Application site discomfort (General disorders) | 1 | 1 | 2
Periorbital oedema (Eye disorders) | 2 | 3 | 2
Eyelid oedema (Eye disorders) | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 3 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Headache (Nervous system disorders) | 1 | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.